CLINICAL TRIAL: NCT05966129
Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics
Brief Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics (Acute Pain Trial)
Acronym: ADOPT PGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); University of Florida (Other); Vanderbilt University Medical Center (Other); Indiana University School of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00104948_A; U01HG010225 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acute Pain
Keywords: Pharmacogenetic; CYP2D6; CYP2C19
MeSH Terms: conditions — Acute Pain | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Immediate vs. delayed pharmacogenetic testing and genotype-guided pain or depression therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Pain - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and clinical decisions support for pain management prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Acute Pain - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing

INTERVENTIONS:
Other: Pharmacogenetic testing — Genetic testing of CYP2D6 and CYP2C19
Other: Clinical decisions support — Prescribing recommendations to the provider based on the pharmacogenetic testing results
  Arms: Acute Pain - Immediate PGx Testing

SUMMARY:
This study is comprised of three separate pharmacogenetic trials grouped into a single protocol due to similarities in the intervention, the hypotheses, and the trial design. The three trials are the Acute Pain Trial, the Chronic Pain Trial, and the Depression Trial. Participants can enroll in only one of the three trials. All three trials were registered on ClinicalTrials.gov under NCT04445792. In July 2023 each of the three treatment trials was registered under a separate NCT# and NCT04445792 was converted to a screening record per recent guidance on master protocol research programs (MPRPs). This record is specific to the Acute Pain Trial within the ADOPT-PGx protocol.

The Acute Pain Trial is a prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided post-surgical opioid therapy (Intervention arm) or standard care and pharmacogenetic testing after 6 months (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype guided pain management therapy improves pain control after surgery in participants who's body processes some pain medicines slower than normal.

DETAILED DESCRIPTION:
Pain and depression are conditions that impact substantial proportions of the US population. Finding safe and effective drug therapies for both conditions is challenging. In the case of treatment for acute and chronic pain, the challenge is finding effective therapy while minimizing adverse effects or opioid addiction (and the ensuing consequences). For depression, there are few clinically relevant predictors of successful treatment leading to multiple trials of inadequate therapy for some patients. Both opioid and antidepressant prescriptions can be guided by pharmacogenetics (PGx) data based on existing guidelines from the Clinical Pharmacogenetics Implementation Consortium (CPIC).

This study is designed to evaluate the impact of pharmacogenetic testing and genotype-guided pain or anti-depressant therapy on pain control or depression symptoms in a pragmatic setting.

The rationale for examining a genotype-guided approach to acute and chronic pain management is based on the importance of CYP2D6 for the bioactivation of tramadol, codeine, and hydrocodone and data from a pilot study supporting improved pain control in intermediate and poor CYP2D6 metabolizers in the genotype-guided arm who are taking these drugs at baseline. Similarly, the rationale for examining a genotype-guided approach to depression medication therapy is based on the demonstrated role of CYP2D6 in the bio inactivation and CYP2C19 oxidation of select, commonly used SSRIs. Secondly, data from industry sponsored trials support the hypothesis of improved depression symptom control in a genotype-guided arm.

Study objectives:

Determine if a genotype-guided approach to acute post-surgical pain therapy leads to improved pain control compared to usual care, as defined by a decrease in the SIA score. Secondarily, The investigators will evaluate whether this approach leads to reduced use of DEA Schedule II opioids and reduced pain intensity.

ELIGIBILITY:
Inclusion Criteria:

Acute Pain Trial

* Age ≥ 8 years
* English speaking or Spanish speaking
* Elective/planned surgery types with planned or anticipated to be treated with tramadol, hydrocodone, or codeine pain management at an enrolling site, which may include orthopedic surgeries (e.g. arthroplasty, spine, etc.), open abdominal surgery, or cardiothoracic surgery and others

Exclusion Criteria

Trial-wide:

* Life expectancy less than 12 months
* Are too cognitively impaired to provide informed consent and/or complete study protocol
* Are institutionalized or too ill to participate (i.e. mental or nursing home facility or incarcerated)
* Have a history of allogeneic stem cell transplant or liver transplant
* People with prior clinical pharmacogenetic test results for genes relevant for the study in which they will enroll (CYP2D6 for the pain studies and CYP2D6 or CYP2C19 for depression) or already enrolled in an ADOPT PGx trial

Acute Pain Trial

* Undergoing a laparoscopic surgery
* Receiving chronic opioid therapy, defined as use of opioids on most days for >3 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1602 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, Study Director — Duke University; Larisa H. Cavallari, PharmD, Principal Investigator — University of Florida; Julie A. Johnson, PharmD, Principal Investigator — Ohio State University
Locations (11):
- United States (11):
  - Nemours Children's Health System, Wilmington, Delaware
  - University of Florida - Gainesville, Gainesville, Florida
  - Nemours Children's Health System, Jacksonville, Florida
  - Nemours Children's Health System, Orlando, Florida
  - Indiana University, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Meharry Medical College, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavallari LH, Cicali E, Wiisanen K, Fillingim RB, Chakraborty H, Myers RA, Blake KV, Asiyanbola B, Baye JF, Bronson WH, Cook KJ, Elwood EN, Gray CF, Gong Y, Hines L, Kannry J, Kucher N, Lynch S, Nguyen KA, Obeng AO, Pratt VM, Prieto HA, Ramos M, Sadeghpour A, Singh R, Rosenman M, Starostik P, Thomas CD, Tillman E, Dexter PR, Horowitz CR, Orlando LA, Peterson JF, Skaar TC, Van Driest SL, Volpi S, Voora D, Parvataneni HK, Johnson JA; IGNITE Pragmatic Trials Network. Implementing a pragmatic clinical trial to tailor opioids for acute pain on behalf of the IGNITE ADOPT PGx investigators. Clin Transl Sci. 2022 Oct;15(10):2479-2492. doi: 10.1111/cts.13376. Epub 2022 Aug 4. PMID 35899435
- See also: Implementing a pragmatic clinical trial to tailor opioids for acute pain on behalf of the IGNITE ADOPT PGx investigators — https://pubmed.ncbi.nlm.nih.gov/35899435/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This record is specific to the Acute Pain Trial within the ADOPT PGx protocol. It only contains the participants consented to the Acute Pain Trial.
Period: Overall Study
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing
Started | 801 | 801
Completed | 645 | 638
Not Completed | 156 | 163
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 63 | 66
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 26 | 25
Not completed — Surgery not completed | 63 | 69
Not completed — Surgery logistics issue | 2 | 1

BASELINE CHARACTERISTICS:
Population: ITT refers to the Intent To Treat population, while mITT, a subset of ITT, refers to the modified Intent To Treat population. The mITT population is the primary analytical population for the Acute Pain Trial defined as participants with a CYP2D6 activity score ≤0.75.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Total
Number analyzed (Participants) | 801 | 801 | 1602
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intent to Treat population
  years | 62.4 (14.2) | 62.8 (13.7) | 62.6 (13.9)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Modified Intent to Treat population
  years
    number analyzed (Participants) | 176 | 175 | 351
    (all) | 62.8 (12.1) | 61.8 (13.1) | 62.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent to Treat population
  Participants
    Female | 494 | 489 | 983
    Male | 307 | 312 | 619
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Modified Intent To Treat population
  Participants
    number analyzed (Participants) | 176 | 175 | 351
    Female | 116 | 122 | 238
    Male | 60 | 53 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat population
  Participants
    Hispanic or Latino | 43 | 54 | 97
    Not Hispanic or Latino | 753 | 739 | 1492
    Unknown or Not Reported | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat population
  Participants
    number analyzed (Participants) | 176 | 175 | 351
    Hispanic or Latino | 5 | 6 | 11
    Not Hispanic or Latino | 170 | 169 | 339
    Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent to Treat population
  Participants
    Race: American Indian or Alaska Native | 3 | 6 | 9
    Race: Asian | 14 | 8 | 22
    Race: Native Hawaiian or Other Pacific Islander | 6 | 2 | 8
    Race: Black or African American | 122 | 104 | 226
    Race: White | 602 | 621 | 1223
    Race: More than one race | 7 | 5 | 12
    Race: Other | 47 | 55 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Modified Intent to Treat population
  Participants
    Race: number analyzed (Participants) | 176 | 175 | 351
    Race: American Indian or Alaska Native | 0 | 3 | 3
    Race: Asian | 8 | 0 | 8
    Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Race: Black or African American | 22 | 29 | 51
    Race: White | 139 | 134 | 273
    Race: More than one race | 0 | 3 | 3
    Race: Other | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 801 | 801 | 1602

OUTCOME MEASURES:

1. Primary Outcome: 10 Day Silverman Integrated Analgesic Assessment (SIA) Score
Description: A composite measure of pain and opioid usage, the Silverman Integrated Analgesic Assessment (SIA) score, at 10 days post-surgery in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75. The SIA has a total score range of -200 to 200, where a higher score corresponds with higher pain and opioid use.
Time Frame: Day of surgery (baseline) to 10 days post surgery
Population: Modified intent to treat (mITT) population, consisting of participants who completed their surgery and have a genotypic or phenoconverted CYP2D6 activity score ≤ 0.75.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT): Immediate genetic testing of CYP2D6 and clinical decisions support for pain management prescribing to the healthcare provider
  Pharmacogenetic testing: Genetic testing of CYP2D6 and CYP2C19
  Clinical decisions support: Prescribing recommendations to the provider based on the pharmacogenetic testing results
- Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT): Delayed genetic testing of CYP2D6 and return of results after the conclusion of the 6-month follow-up period
  Pharmacogenetic testing: Genetic testing of CYP2D6 and CYP2C19
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 160 | 152
score on a scale | 1.4 (95.9) | -1.4 (93.1)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.7957, t-test, 2 sided; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-18.3 to 23.8]; Confidence Interval Width = 42.1

2. Secondary Outcome: 10 Day Pain Intensity as Measured by the PROMIS Numeric Pain Rating Scale
Description: PROMIS (Patient-Reported Outcomes Measurement Information System) Numeric Pain Rating Scale Pain intensity at 10 days post-surgery in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75. Pain was measured on a scale of 0-10, where higher scores correspond to higher levels of pain.
Time Frame: 10 days post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 168 | 160
score on a scale | 5.2 (2.2) | 5.1 (2.3)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.8255, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.5]; Confidence Interval Width = 0.9

3. Secondary Outcome: Post-surgery Opioid Usage, Measured in Milligrams of Morphine Equivalents (MME) Per Day
Description: Opioid usage from surgery to 10 days post-surgery in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75.
Time Frame: Day of surgery (baseline) to 10 days post surgery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: MME/day
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 160 | 152
MME/day | 10.0 [3.0 to 20.0] | 8.9 [3.5 to 18.4]
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.9054, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: 3 Month Prescription Pain Medication Misuse
Description: The 7-item PROMIS Prescription Pain Medication Misuse questionnaire assesses the extent to which participants experience medication misuse symptoms over the past 3 months using a 5-point Likert scale. The 7 questions are converted to a raw score, ranging from 7 to 35. Raw scores are converted to T-scores using the PROMIS conversion tables and range from 36.3 to 55.8. Higher scores reflect greater medication misuse.
Time Frame: 3 months post surgery
Population: Modified intent to treat (mITT) population, consisting of participants who completed their surgery and have a genotypic or phenoconverted CYP2D6 activity score ≤ 0.75 who indicated having a prescription for pain medication in the past 3 months.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 93 | 98
T-score | 38.5 (3.8) | 39.2 (4.5)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.248, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.9 to 0.5]; Confidence Interval Width = 2.4

5. Secondary Outcome: 1 Month PROMIS Mobility Score
Description: PROMIS mobility score at 1 month post-surgery in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75 in the adult population only. The score ranges from 15 to 75, where a higher score corresponds to higher mobility.
Time Frame: 1 month post surgery
Population: Modified intent to treat (mITT) population, consisting of participants who completed their surgery and have a genotypic or phenoconverted CYP2D6 activity score ≤ 0.75 in adults only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 164 | 161
score on a scale | 40.4 (16.6) | 39.4 (17.2)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.6012, t-test, 2 sided; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-2.7 to 4.7]; Confidence Interval Width = 7.4

6. Secondary Outcome: Number of Participants With Opioid Persistence
Description: Opioid persistence defined as a filled prescription for an opioid medication 3-6 months post-surgery in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75.
Time Frame: 3-6 months post-surgery, assessed at 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 153 | 146
Participants | 24 | 21
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p = 0.7528, Chi-squared

7. Secondary Outcome: Participants With Drug-Gene Concordance
Description: Drug-Gene Concordance defined as an agreement between the Pharmacogenomics (PGx) Test and the prescribed opioids post surgery for pain management in participants who have a genotypic or pheno-converted CYP2D6 activity score ≤ 0.75
Time Frame: Within 10 days post-surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) | Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT)
Number analyzed (Participants) | 176 | 175
Participants | 112 | 47
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing (Modified Intent-to-treat, mITT) vs Acute Pain - Delayed PGx Testing (Modified Intent-to-treat, mITT); Test type: Superiority; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Per the study protocol, only Adverse Device Effect (ADE) events suspected to be related to the specimen collection, laboratory assay genotyping results, and phenoconversion recommendations from the Best Practice Alerts (BPAs)/Consult notes were collected.
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing
All-Cause Mortality (participants affected / at risk) | 1/801 | 2/801
Serious Adverse Events (participants affected / at risk) | 0/801 | 0/801
Other Adverse Events (participants affected / at risk) | 0/801 | 0/801

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05966129/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT05966129/ICF_000.pdf